CLINICAL TRIAL: NCT07024173
Title: A Multicenter, Open-label, Randomized Controlled Phase 3 Study of HRS-8080 Versus Treatment Chosen by Physicians in Locally Advanced and Metastatic Breast Cancer With Disease Progression After Previous Endocrine Therapy
Brief Title: A Phase 3 Study of HRS-8080 Versus Treatment Chosen by Physicians in Locally Advanced and Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-8080-303
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; exemestane; Everolimus; Anastrozole; Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HRS-8080 Group (Experimental)
  Interventions: Drug: HRS-8080 Tablet
- Fulvestrant Group (Active Comparator)
  Interventions: Drug: Fulvestrant injection
- Exemestane in combination with Everolimus Group (Active Comparator)
  Interventions: Drug: Exemestane tablets; Drug: Everolimus Tablets
- Exemestane or Anastrozole or Letrozole Group (Active Comparator)
  Interventions: Drug: Exemestane tablets; Drug: Anastrozole Tablets; Drug: Letrozole Tablets

INTERVENTIONS:
Drug: HRS-8080 Tablet — HRS-8080 tablet orally administered.
  Arms: HRS-8080 Group
Drug: Fulvestrant injection — Fulvestrant injection.
  Arms: Fulvestrant Group
Drug: Exemestane tablets — Exemestane tablets orally administered.
  Arms: Exemestane in combination with Everolimus Group; Exemestane or Anastrozole or Letrozole Group
Drug: Everolimus Tablets — Everolimus tablets orally administered.
  Arms: Exemestane in combination with Everolimus Group
Drug: Anastrozole Tablets — Anastrozole tablets orally administered.
  Arms: Exemestane or Anastrozole or Letrozole Group
Drug: Letrozole Tablets — Letrozole tablets orally administered.
  Arms: Exemestane or Anastrozole or Letrozole Group

SUMMARY:
This study is a multicenter, open-label, randomized controlled Phase 3 clinical trial. It is planned to enroll 240 female patients with locally advanced or metastatic breast cancer followed by disease progression after previous endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 to 75 years old (including both values).
2. ECOG Physical Strength Status (PS) : 0 to 1 point.
3. Patients with locally advanced or metastatic breast cancer confirmed by histology.
4. Patients previously received 1-2 lines of endocrine therapy.
5. Expected survival > 6 months.
6. The functional level of the organs must meet the requirements.
7. Subjects that voluntarily participate in this clinical trial, be willing and able to abide by the procedures related to clinical visits and research, understand the research procedures and have signed the informed consent.

Exclusion Criteria:

1. Patients with rapid disease progress and investigators determine that endocrine therapy is not suitable or tolerant.
2. A history of severe clinical cardiovascular diseases.
3. Patients with uncontrollable tumor-related pain as judged by investigators.
4. Severe infection exists within 4 weeks before the first study administration.
5. Patients with clinically significant endometrial abnormalities.
6. Untreated active hepatitis.
7. Patients known to be allergic to HRS-8080 components.
8. Pregnant and lactating women, or those planning to become pregnant during the study period.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) evaluated by the blinded independent central review (BICR). | Approximately 2 years.

SECONDARY OUTCOMES:
Progression free survival (PFS) evaluated by investigators. | Approximately 2 years.
Overall response rate (ORR). | Approximately 2 years.
Clinical benefit rate (CBR). | Approximately 2 years.
Duration of response (DOR). | Approximately 2 years.
Overall survival (OS). | Approximately 3 years.
Adverse events (AEs). | Approximately 2 years.
Serious adverse events (SAEs). | Approximately 2 years.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: Undecided